CLINICAL TRIAL: NCT02201498
Title: A New Technique for Primary Molar Pulpotomy : A Randomized Clinical Trial Comparing the Radiographic and Clinical Success of the Formocresol-zinc Oxide Eugenol Technique and the Biodentine Technique
Brief Title: Randomized Clinical Trial for Primary Molar Pulpotomy, Biodentine Vs Formocresol-ZOE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Montréal (Other)
Collaborators: Septodont (Industry); St. Justine's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BIODENT1
Record Dates: First submitted 2014-07-24; First posted 2014-07-28 (Estimated); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Deep Dental Caries
MeSH Terms: interventions — Pulpotomy; tricalcium silicate

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Formocresol/OZE (Active Comparator): Conventional pulpotomy technique, with formocresol and zinc oxide eugenol
  Interventions: Procedure: Pulpotomies with Formocresol/OZE and Biodentine
- Biodentine (Active Comparator): New technique, with biodentine
  Interventions: Procedure: Pulpotomies with Formocresol/OZE and Biodentine

INTERVENTIONS:
Procedure: Pulpotomies with Formocresol/OZE and Biodentine

SUMMARY:
This is a RCT that will compare the clinical and radiographic success of pulpotomies on primary molars between the traditional technique (Formocresol/ZOE) and the new technique with Biodentine. 180 pulpotomies (90 in each group) will be followed for a period of 12 months.

ELIGIBILITY:
Inclusion Criteria:

* ASA I and II
* less than 1/3 of physiologic root resorption
* asymptomatic tooth (with no history of symptoms)
* no clinical or radiological sign of pathology
* vital tooth, with carious pulpal exposure
* hemostasis must be obtained simply with pressure in less than 5 min
* teeth restored with stainless steel crowns

Exclusion Criteria:

* more than 10 y.o.
* symptomatic tooth (presently or history of symptoms)
* previous pulpal treatment on the tooth
* necrotic pulp
* hyperemic pulp
* inadequate operative technique, defective restauration
* non diagnostic x-ray (pre or post treatment)

Max Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
clinical success | 12 months post treatment
radiographic success | 12 months post treatment

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Sainte-Justine, Montreal, Quebec, Canada